CLINICAL TRIAL: NCT03020368
Title: Effectiveness and Safety of Breeded Leech "Medileech" by BioRepro GmbH for Symptomatic Primary Arthrosis of the First Carpometacarpal Joint: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness and Safety of Breeded Leech for Symptomatic Primary Arthrosis of the First Carpometacarpal Joint
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Leeches for Rhizarthrosis
Record Dates: First submitted 2017-01-11; First posted 2017-01-13 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Rhizarthrosis
MeSH Terms: interventions — Leeching; Diclofenac

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Leeches (Experimental): One-time topical application of 2-3 leeches ("medileech", Hirudo verbana) periarticularly on the painful thumb base
  Interventions: Biological: Leeches
- Diclofenac (Active Comparator): 3 times daily topical application of Diclofenac gel (1 g with 10 mg diclofenac-Na) over 4 weeks
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Biological: Leeches
  Other Names: Hirudo verbana
  Arms: Leeches
Drug: Diclofenac
  Arms: Diclofenac

SUMMARY:
In this trial the investigators want to prove the efficacy and safety of a one-time topical leech application at patients with symptomatic primary arthrosis of the first carpometacarpal joint in comparison to the standard therapy with topical diclofenac.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 35 to 85 years
* Pain intensity in the region of the thumb base in pain phases ≥ 40 mm on the VAS of 0 to 100 mm (relative to the last 24 hours)
* Complaints for at least 3 months
* X-ray Stadium Eaton I-IV at least once secured

Exclusion Criteria:

* Anticoagulation (Marcumar, Heparin)
* Haemophilia, V. Willebrandt Jürgens syndrome, thrombocytopathy and other blood anomalies
* Combination therapy of ASA and thienopyridines
* Pain medication with opioid analgesics
* Systemic medication with corticoids or immunosuppressants
* Intraarterticular injections or RSO within the last 3 months
* Past or planned surgery on the affected joint in the next 2 months
* Pregnancy, lactation
* Insulin-dependent type I diabetes mellitus
* Acute psychotic disorders
* Severe comorbidity

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | Change after 28 and 56 days

SECONDARY OUTCOMES:
Visual analog scale (VAS) | Change after 7, 28 and 56 days
Medication on demand | Documentation between baseline and day 56
  Documentation in daily diary

OTHER OUTCOMES:
Expectation | Baseline
  5-stage Likert scale for the expectation of symptomatic efficacy after group assignment
Overall assessment of efficacy and tolerability | Day 56
  5-stage Likert scale documented by the patient as well as by the doctor at the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, Prof. Dr., Principal Investigator — Charite Centrum Epidemiologie und Gesundheitsökonomie, CC1: Gesundheitswissenschaften
Locations (1):
- Hochschulambulanz für Naturheilkunde der Charité-Universitätsmedizin Berlin am Immanuel-Krankenhaus, Berlin, Germany